CLINICAL TRIAL: NCT02760641
Title: Does an Egg-Rich Diet Improve Metabolic Health and Function in Obese Older Adults
Brief Title: Egg Diet to Improve Metabolic Health and Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: American Egg Board (Other)
Responsible Party: Principal Investigator, Kevin Fontaine, Principal Investigators, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F141016101
Record Dates: First submitted 2016-04-28; First posted 2016-05-03 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2016-10

CONDITIONS: Obesity
Keywords: obesity; low carbohydrate diet; metabolism; body composition; visceral fat; older adults; insulin sensitivity
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Egg-based diet (EBD) (Experimental): This arm will provide ≤25% energy from CHO, 25% energy from protein, and ≥50% energy from fat. EBD participants will be asked to consume ≥2 eggs per day along with other protein sources including meat, fish, pork, and poultry. Carbohydrate (CHO) sources will be primarily derived from leafy greens and non-starchy vegetables and CHO intake will be equally distributed across meals throughout the day.
  Interventions: Other: Egg-based diet (EBD)
- Carbohydrate-based diet (CBD) (Placebo Comparator): The CBD group will be asked to avoid whole egg consumption when possible during the 8 week intervention period. They will be counseled to consume a low fat diet with 55:25:20 %energy from CHO:protein:fat. This diet will place an emphasis on consuming lean meats, low fat dairy, whole grains, legumes, fruits and vegetables.
  Interventions: Other: Carbohydrate-based diet (CBD)

INTERVENTIONS:
Other: Egg-based diet (EBD) — Participants will be asked to consume a carbohydrate-restricted diet including whole eggs for 8 weeks. Eggs will be provided.
  Arms: Egg-based diet (EBD)
Other: Carbohydrate-based diet (CBD) — Participants will be asked to consume a low fat, carbohydrate-based diet for 8 weeks. Breakfast food items will be provided.
  Arms: Carbohydrate-based diet (CBD)

SUMMARY:
The purpose of this study is to determine the effects of change in diet quality (carbohydrate restriction versus fat restriction) on body composition, fat distribution, cardiometabolic risk factors, physical function, and quality of life in aging adults with obesity.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effects of change in diet quality (carbohydrate restriction versus fat restriction) on body composition, fat distribution, cardiometabolic risk factors, physical function, and quality of life in aging adults with obesity. Data from previous studies support the hypothesis that consumption of lower-CHO, higher-fat food sources rich in high-quality proteins and essential fatty acids, such as whole eggs, has beneficial effects on metabolic health. The study will test the hypothesis that a reduced CHO higher- fat, egg-rich diet induces selective depletion of total and abdominal adiposity, preserves lean mass, and reduces inflammation and oxidative stress. In turn, these favorable changes in body composition, fat distribution, and metabolic health will confer improvements in physical function in obese, aging adults.

Results from this study will form an empirical basis for developing an easily implemented, non-pharmacologic treatment (i.e. change diet quality by incorporating more low carbohydrate, whole foods such as eggs) to prevent or reverse sarcopenia and other age-related diseases of metabolic origins.

ELIGIBILITY:
Inclusion Criteria:

1. between 60-75 years of age,
2. have a BMI ranging from 30-40 kg/m2,
3. sedentary (<2h/wk of intentional exercise, and agree to maintain their level of activity throughout the study).

Exclusion Criteria:

1. those with uncontrolled diabetes,
2. unwilling to eat the prescribed diets,
3. recent weight change (+/- 10 lbs. in previous year),
4. history of eating disorder,
5. difficulty chewing and swallowing solid food,
6. digestive diseases,
7. cognitive impairment,
8. uncontrolled blood pressure (systolic blood pressure > 159 or diastolic blood pressure >95 mm Hg),
9. history of non-skin cancer in the last 5 years,
10. cardiovascular disease event; severe pulmonary disease; renal failure; major liver dysfunction,
11. current/recent smoker,
12. use of estrogen or testosterone replacement therapy,
13. current use of oral corticosteroids (>5 d/mth),
14. using medications for treatment of psychosis or manic-depressive illness, and
15. dependence on others for food procurement or preparation.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-01; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Changes in total fat mass as measured by dual-energy X-ray absorptiometry (DXA) | 8 weeks after baseline
Changes in visceral adipose tissue as measured by magnetic resonance imaging (MRI) | 8 weeks after baseline
Changes in total lean mass as measured by DXA | 8 weeks after baseline
Changes in subcutaneous abdominal adipose tissue as measured by MRI | 8 weeks after baseline
Changes in thigh intermuscular adipose tissue as measured by MRI | 8 weeks after baseline
Changes in thigh skeletal muscle volume as measured by MRI | 8 weeks after baseline
Changes in thigh subcutaneous adipose tissue as measured by MRI | 8 weeks after baseline

SECONDARY OUTCOMES:
Changes in pro-inflammatory markers, Interleukin (IL)-6 | 8 weeks after baseline
Changes in pro-inflammatory marker, hsCRP | 8 weeks after baseline
Changes in pro-inflammatory marker, Tumor Necrosis Factor (TNF)-α | 8 weeks after baseline
Changes in metabolic hormone adiponectin | 8 weeks after baseline
Changes in metabolic hormone leptin | 8 weeks after baseline
Changes in metabolic hormone insulin | 8 weeks after baseline
Changes in markers of oxidative stress : isoprostanes | 8 weeks after baseline
Changes in markers of oxidative stress : protein carbonyls | 8 weeks after baseline
Changes in markers of oxidative stress : total anti-oxidants | 8 weeks after baseline
Changes in insulin sensitivity with euglycemic-hyperinsulinemic clamp | 8 weeks after baseline
Changes in the lipid profile: triglycerides | 8 weeks after baseline
Changes in the lipid profile: total cholesterol | 8 weeks after baseline
Changes in the lipid profile: HDL-C | 8 weeks after baseline
Changes in the lipid profile: LDL | 8 weeks after baseline
Changes in physical function: Short Physical Performance Battery | 8 weeks after baseline
Changes in physical function : muscle strength | 8 weeks after baseline
Changes in quality of life (SF-36 Health Survey). | 8 weeks after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Kevin M Fontaine, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hoover SE, Il'yasova D, Fontaine KR, Spasojevic I, Gower BA, Goss AM. A Pilot Study of Associations Between Visceral Fat, IL-6, and Urinary F2-Isoprostanes in Older Adults Exposed to a Diet Intervention. Curr Dev Nutr. 2021 May 21;5(6):nzab082. doi: 10.1093/cdn/nzab082. eCollection 2021 Jun. PMID 34212125
- [Derived] Goss AM, Gower B, Soleymani T, Stewart M, Pendergrass M, Lockhart M, Krantz O, Dowla S, Bush N, Garr Barry V, Fontaine KR. Effects of weight loss during a very low carbohydrate diet on specific adipose tissue depots and insulin sensitivity in older adults with obesity: a randomized clinical trial. Nutr Metab (Lond). 2020 Aug 12;17:64. doi: 10.1186/s12986-020-00481-9. eCollection 2020. PMID 32817749